CLINICAL TRIAL: NCT02875145
Title: Impact of Cataract Surgery on Keratoplasty Graft Survival
Acronym: IGREC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: API/2014/53
Record Dates: First submitted 2016-07-28; First posted 2016-08-23 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Cataract; Fuchs' Endothelial Dystrophy; Keratoconus
Keywords: Corneal Transplantation; Graft Survival
MeSH Terms: conditions — Cataract; Fuchs' Endothelial Dystrophy; Keratoconus | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Keratoplasty with cataract surgery: Patients who underwent keratoplasty who also underwent a cataract surgery during follow up.
  Interventions: Procedure: Cataract surgery
- Keratoplasty without cataract surgery: Patients who underwent keratoplasty who never underwent cataract surgery.

INTERVENTIONS:
Procedure: Cataract surgery
  Groups: Keratoplasty with cataract surgery

SUMMARY:
The follow up time after keratoplasty now routinely exceeds multiple decades. It is common for keratoplasty patients to also undergo cataract surgery at a later date in their lives.

Keratoplasties and cataract surgery both result in local inflammation. This may influence the density of endothelial cells, and on average there is a loss of 10% in endothelial cells within 3 months of the cataract surgery. Yet, a sufficient density of endothelial cells is required to maintain graft transparency. It may be therefore difficult to strike a balance between loss of visual acuity due to the cataract of to the loss of graft transparency over the long term.

The investigators aim to compare graft survival in patients with clear crystalline lens with and without cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing keratoplasty
* Between january 1983 and december 2012
* Age 40 and older at the time of surgery

Exclusion Criteria:

* Cataract surgery prior to the keratoplasty
* Systemic inflammatory disease
* Previous history of uveitis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent a keratoplasty between january 1983 and december 2012 at the University Hospital of Besançon.
Sampling Method: Non-Probability Sample
Enrollment: 453 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Corneal transplant graft survival | 10 years

SECONDARY OUTCOMES:
Corneal endothelial cell density | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Delbosc, MD, PhD, Principal Investigator — Opthalmology Department, CHU Besançon
Locations (1):
- Ophthalmology Department, CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No